CLINICAL TRIAL: NCT00331513
Title: A Phase 1 Study of Suberoylanilide Hydroxamic Acid (Vorinostat, SAHA) in Combination With Idarubicin in Relapsed or Refractory Leukemia
Brief Title: Vorinostat and Idarubicin in Treating Patients With Relapsed or Refractory Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00094; NCI-2009-00094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000472062; 2005-0031 (Other: M D Anderson Cancer Center); 6892 (Other: CTEP); U01CA062461 (NIH)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Promyelocytic Leukemia (M3); Blastic Phase Chronic Myelogenous Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Promyelocytic, Acute; Blast Crisis; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Vorinostat; Idarubicin

ARMS (2):
- Arm I (vorinostat, idarubicin) (Active Comparator): Patients receive oral SAHA three times daily on days 1-14 and idarubicin IV over 15 minutes once daily on days 1-3. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients completing 6 courses of therapy or who reach the maximum cumulative dose of idarubicin or an equivalent anthracycline and achieve clinical benefit may continue treatment with SAHA alone 3 times daily on days 1-14 of each course, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: idarubicin; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (vorinostat, idarubicin) (Active Comparator): Patients receive oral SAHA three times daily and idarubicin IV over 15 minutes once daily on days 1-3. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients completing 6 courses of therapy or who reach the maximum cumulative dose of idarubicin or an equivalent anthracycline and achieve clinical benefit may continue treatment with SAHA alone 3 times daily on days 1-14 of each course, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: idarubicin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of vorinostat when given together with idarubicin in treating patients with relapsed or refractory leukemia or myelodysplastic syndromes. Drugs used in chemotherapy, such as vorinostat and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with idarubicin may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicities of vorinostat (SAHA) in combination with standard-dose idarubicin in patients with relapsed or refractory acute myeloid leukemia, acute lymphocytic leukemia, myelodysplastic syndromes, acute promyelocytic leukemia, or chronic myelogenous leukemia in blastic phase.

II. Describe the clinical activity of this regimen in these patients. III. Determine the in vivo molecular effects of this regimen, including the effects on DNA topoisomerase IIα mRNA expression and on the induction of γH2AX, histone H3 and H4 acetylation, as well as changes in the gene expression profile.

IV. Determine the pharmacokinetic characteristics of this regimen in these patients.

OUTLINE:

This is a randomized, dose-escalation study of vorinostat (SAHA). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral SAHA three times daily on days 1-14 and idarubicin IV over 15 minutes once daily on days 1-3. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.*

ARM II: Patients receive oral SAHA three times daily and idarubicin IV over 15 minutes once daily on days 1-3. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.*

Note: *Patients completing 6 courses of therapy or who reach the maximum cumulative dose of idarubicin or an equivalent anthracycline and achieve clinical benefit may continue treatment with SAHA alone 3 times daily on days 1-14 of each course, in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience a dose-limiting toxicity. An additional 10 patients are treated at the MTD.

Patients undergo blood collection and bone marrow biopsies periodically during the study for pharmacologic, biomarker, and genetic studies.

After completion of study treatment, patients are followed at 4 weeks and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed/refractory acute myelogenous leukemia, acute lymphocytic leukemia, myelodysplastic syndrome or blastic phase chronic myelogenous leukemia.
* Patients that have received cumulative doses (or its equivalent to other anthracycline) of more than 290 mg/m^2 of idarubicin will be excluded from the study. No other limitations in terms of number of prior therapies or type of therapies apply to this study.
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Total bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 2 mg/dL
* LVEF ≥ 50%
* Not nursing or pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 2 weeks since prior chemotherapy and recovered, unless there is evidence of rapidly progressive disease, at least 24 hours since prior hydroxyurea for rapidly proliferating disease
* At least 2 weeks since prior imatinib mesylate
* At least 2 weeks since prior histone deacetylase inhibitors, including valproic acid
* Maximum cumulative dose of prior idarubicin or equivalent anthracycline drug ≤ 290 mg/m2
* No concurrent epoetin alfa or hematopoietic colony-stimulating factors during the first course of study therapy
* No concurrent prophylactic hematopoietic colony-stimulating factors
* Myelodysplastic syndromes requiring treatment, previously treated with either azacytidine or decitabine, unless it was contraindicated; blastic phase chronic myelogenous leukemia; failed prior imatinib mesylate-based therapy
* Patients with MDS should have received therapy with either 5-azacytidine or 5-aza-2'-deoxycytidine, unless the patient had a contraindication to such therapy, and should require therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with clinical evidence of CNS disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* No unstable angina pectoris
* Considered ineligible for or refused potentially curative therapy, including allogeneic stem cell transplantation, with or without standard induction therapy
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to vorinostat (SAHA) or other agents used in this study
* No ongoing or active infection
* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of vorinostat determined by dose-limiting toxicities (DLT) as measured by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.3.0 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States